CLINICAL TRIAL: NCT01316146
Title: Phase I Study of the Administration of T Lymphocytes Expressing the CD30 Chimeric Antigen Receptor for Relapsed CD30+ Hodgkin's Lymphoma and CD30+ Non-Hodgkin's Lymphoma (CART CD30)
Brief Title: Administration of T Lymphocytes for Hodgkin's Lymphoma and Non-Hodgkin's Lymphoma (CART CD30)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never truly opened to accrual at UNC. Study and data were transfered to UNC as the IND for the study was transfered to UNC. IRB closed the study.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Baylor College of Medicine (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1544-ATL; H-27721-CART CD30 (Other: Baylor)
Record Dates: First submitted 2011-03-04; First posted 2011-03-16 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Lymphoma; T lymphocytes
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAR.CD30 T cells (Experimental): Three dose levels will be evaluated. Using the modified continual reassessment method, cohorts of size two will be enrolled at each dose level. Each patient will receive one injection (IV) according to the dosing schedules: starting with the lowest cell dose (2×10^7 cells/m2) and then escalate the cell dose to the highest cell dose (2×10^8/m2) as per study design.
  Interventions: Drug: CAR.CD30 T cells

INTERVENTIONS:
Drug: CAR.CD30 T cells — Three dose levels will be evaluated:
  Group One, 2x10^7 cells/m^2
  Group Two, 1x10^8 cells/m^2
  Group Three, 2x10^8 cells/m^2;
  Cell Administration: CAR+ ATL will be given by intravenous injection over 1-10 minutes through either a peripheral or a central line. The expected volume will be 1-50cc.

SUMMARY:
The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancer. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from diseases caused by germs or toxic substances. They work by binding those germs or substances, which stops them from growing and causing bad effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected with germs. Both antibodies and T cells have been used to treat patients with cancers: they both have shown promise, but have not been strong enough to cure most patients. Investigators hope that both will work better together.

Investigators have found from previous research that they can put a new gene into T cells that will make them recognize cancer cells and kill them. Investigators now want to see if they can attach a gene to T cells that will help them do a better job at recognizing and killing lymphoma cells.

The new gene that investigators will put in T cells makes an antibody called anti-CD30. This antibody sticks to lymphoma cells because of a substance on the outside of the cells called CD30. Anti-CD30 antibodies have been used to treat people with lymphoma, but have not been strong enough to cure most patients.

For this study, the anti-CD30 antibody has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way, it is called a chimeric receptor. These CD30 chimeric receptor-activated T cells seem to kill some of the tumor, but they don't last very long and so their chances of fighting the cancer are unknown.

DETAILED DESCRIPTION:
When the patient enrolls on this study, they will be assigned a dose of CD30 chimeric receptor-activated T cells. The dose level of cells that they will receive will not be based on a medical determination of what is best for the patient, instead the dose is based on the order in which the patient enrolled on the study relative to other participants. Subjects enrolled earlier in the study will receive a lower dose of cells than those enrolled later in the study. The risks of harm and discomfort from the study treatment may bear some relationship to the dose level. The potential for direct benefit, if any, may also vary with the dose level.

The patient will be given an injection of CD30 chimeric receptor-activated T cells into the vein through an IV line at the assigned dose. The injection will take 1-10 minutes. Investigators will follow the subject in the clinic after the injection for up to 4 hours.

To learn more about the way the CD30 chimeric receptor-activated T cells are working and how long they last in the body, extra blood will be drawn.

If the patient has stable disease (the lymphoma did not grow) or there is a reduction in the size of the lymphoma on imaging studies after the T-cell infusion, s/he can receive up to six additional doses of the T cells at 8 to 12 weeks intervals if s/he wishes. After each T-cell infusion, s/he will be monitored as described above.

ELIGIBILITY:
INCLUSION CRITERIA

Procurement Inclusion Criteria:

Referred patients will initially be consented for procurement of blood for generation of the transduced ATL. Eligibility criteria at this stage include:

* Diagnosis of recurrent CD30+ HL or CD30+ NHL, or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of relapsed/refractory CD30+ HL or CD30+ NHL with a treatment plan that will include high dose therapy and stem cell transplantation
* CD30 positive tumor (result can be pending at this time)
* Hgb > 8.0
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.
* Karnofsky or Lansky score greater than 60%

Procurement Exclusion Criteria

- Active infection with HIV, HTLV, HBV, HCV (can be pending at this time).

Treatment Inclusion Criteria:

Diagnosis - CD30+ HL or CD30+ NHL:

1. During the Dose Escalation Phase: only adult patients with active disease failing standard therapy
2. After Dose Escalation: any patient (children or adults) newly diagnosed, unable to receive or complete standard therapy OR diagnosis of relapsed/refractory CD30+ HL or CD30+ NHL with a treatment plan that will include high dose therapy and autologous stem cell transplantation. (During dose escalation: only adult patients (age 18 and older; After Dose Escalation: any patient (children ages 0-17 or adults)

   * CD30 positive tumor
   * Bilirubin 1.5 times or less than upper limit of normal.
   * AST 3 times or less than upper limit of normal.
   * Serum creatinine 1.5 times or less than upper limit of normal.
   * Pulse oximetry of > 90% on room air
   * Karnofsky or Lansky score of > 60%.
   * Available autologous T cells with 15% or more expression of CD30CAR determined by flow-cytometry.
   * Recovered from acute toxic effects of all prior chemotherapy at least one week and 30 days from prior chemotherapy before entering this study
   * Adequate pulmonary function with FEV1, FVC and DLCO greater than or equal to 50% of expected corrected for hemoglobin.
   * Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
   * Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

EXCLUSION CRITERIA:

Procurement Exclusion Criteria:

- Active infection with HIV, HTLV, HBV, HCV (can be pending at this time).

Treatment Exclusion Criteria:

* Currently receiving any investigational agents or received any tumor vaccines within the previous six weeks.
* Received anti-CD30 antibody-based therapy within the previous 4 weeks.
* History of hypersensitivity reactions to murine protein-containing products.
* Pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction.
* Current use of systemic corticosteroids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10-03 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of escalating doses of autologous activated T lymphocytes | 6 weeks
  To evaluate the safety of escalating doses of autologous activated T lymphocytes (ATL), genetically modified to express an artificial chimeric antigen receptor (CAR) that targets the CD30 molecule (CAR.CD30) and also contains the CD28 endodomain, in patients with CD30+ refractory/relapsed Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL).

SECONDARY OUTCOMES:
Measure the survival of CAR.CD30 in vivo | 15 years
  To measure the survival of CAR.CD30 transduced ATL in vivo.
Measure the response of the subjects tumor to the CAR.CD30 transduced ATL | 15 years
  To measure the anti-tumor effects of CAR.CD30 transduced ATL in patients with CD30+ refractory/relapsed Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Savoldo, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos CA, Ballard B, Zhang H, Dakhova O, Gee AP, Mei Z, Bilgi M, Wu MF, Liu H, Grilley B, Bollard CM, Chang BH, Rooney CM, Brenner MK, Heslop HE, Dotti G, Savoldo B. Clinical and immunological responses after CD30-specific chimeric antigen receptor-redirected lymphocytes. J Clin Invest. 2017 Sep 1;127(9):3462-3471. doi: 10.1172/JCI94306. Epub 2017 Aug 14. PMID 28805662